CLINICAL TRIAL: NCT01890317
Title: Randomized Pilot Study of Mild Hypothermia in Cardiogenic Shock Complicating Myocardial Infarction
Brief Title: Mild Hypothermia in Cardiogenic Shock Complicating Myocardial Infarction
Acronym: SHOCK-COOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Holger Thiele, Co-Director Clinic for Internal Medicine/Cardiology, Heart Center Leipzig - University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HZLCOOL1
Record Dates: First submitted 2013-06-24; First posted 2013-07-01 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Acute; Myocardial Infarction, Complications; Cardiogenic Shock
Keywords: Cardiogenic shock; acute myocardial infarction; mild hypothermia
MeSH Terms: conditions — Myocardial Infarction; Shock, Cardiogenic | interventions — Hypothermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mild hypothermia (Experimental): Induction of mild hypothermia for 24 hr with invasive cooling in addition to primary percutaneous coronary intervention and optimal medical therapy
  Interventions: Procedure: Mild hypothermia
- Control (No Intervention): Percutaneous coronary intervention and optimal medical therapy according to current guidelines

INTERVENTIONS:
Procedure: Mild hypothermia — Induction of mild hypothermia with invasive cooling for 24 hr in addition to primary percutaneous coronary intervention and optimal medical therapy.
  Arms: Mild hypothermia

SUMMARY:
Prospective, randomized, single-center, controlled, open-label Pilot-study to investigate whether induction of mild hypothermia in addition to primary percutaneous coronary intervention and optimal medical therapy in myocardial infarction complicated by cardiogenic shock improves cardiac power index after 24 h.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction complicated by cardiongenic shock
* Patients on mechanical ventilation at time of randomization

Exclusion Criteria:

* Out of hospital resuscitation with indication for mild hypothermia
* mechanical complications after acute myocardial infarction
* duration of cardiogenic shock > 12 hours
* age > 90 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Cardiac Power Index after 24 hr. | 24 hours
  Cardiac Power Index after 24 hours as surrogate endpoint.

SECONDARY OUTCOMES:
30-days mortality | 30 days
Change of hemodynamics over the first 48 hr. | During first 48 hr
Catecholamine dose and duration of catecholamine support | 30 days
Length of ICU-stay | 30 days
Length of mechanical ventilation | 30 days
SAPS-II-Score | 96 hours
  Simplified Acute Physiology Score for the first 4 days
Severe and moderate bleeding complications (GUSTO-definition) | 30 days
Sepsis | 30 days
Pneumonia | 30 days
Stroke | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, MD, Study Chair — Heart Center Leipzig - University Hospital; Georg Fuernau, MD, Principal Investigator — Heart Center Leipzig - University Hospital
Locations (1):
- Department of Internal Medicine/Cardiology, University of Leipzig - Heart Center, Leipzig, Saxony, Germany

REFERENCES:
- [Derived] Cheng W, Fuernau G, Desch S, Freund A, Feistritzer HJ, Poss J, Buettner P, Thiele H. Circulating Monocyte Chemoattractant Protein-1 in Patients with Cardiogenic Shock Complicating Acute Myocardial Infarction Treated with Mild Hypothermia: A Biomarker Substudy of SHOCK-COOL Trial. J Cardiovasc Dev Dis. 2022 Aug 20;9(8):280. doi: 10.3390/jcdd9080280. PMID 36005444
- [Derived] Fuernau G, Beck J, Desch S, Eitel I, Jung C, Erbs S, Mangner N, Lurz P, Fengler K, Jobs A, Vonthein R, de Waha-Thiele S, Sandri M, Schuler G, Thiele H. Mild Hypothermia in Cardiogenic Shock Complicating Myocardial Infarction. Circulation. 2019 Jan 22;139(4):448-457. doi: 10.1161/CIRCULATIONAHA.117.032722. PMID 30026282